CLINICAL TRIAL: NCT00216060
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled Trial Evaluating the Ability of Risedronate to Prevent Skeletal Related Events in Patients With Metastatic Prostate Cancer Commencing Hormonal Therapy: Hoosier Oncology Group GU02-41
Brief Title: Risedronate to Prevent Skeletal Related Events in Patients With Metastatic Prostate Cancer Commencing Hormonal Therapy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Terminated due to low accrual
Sponsor: Christopher Sweeney, MBBS (Other)
Collaborators: Sanofi (Industry); Walther Cancer Institute (Other); Hoosier Cancer Research Network (Other)
Responsible Party: Sponsor-Investigator, Christopher Sweeney, MBBS, Sponsor-Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HOG GU02-41
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Results first posted 2016-05-26 (Estimated); Last update posted 2016-05-26 (Estimated); Status verified 2016-05

CONDITIONS: Metastatic Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Risedronic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental Arm (Experimental): Daily oral risedronate combined with androgen deprivation
  Interventions: Drug: Risedronate
- Placebo Arm (Placebo Comparator): daily oral placebo combined with androgen deprivation
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Risedronate — Daily oral risedronate combined with androgen deprivation
  Arms: Experimental Arm
Drug: Placebo — Daily oral placebo combined with androgen deprivation
  Arms: Placebo Arm

SUMMARY:
Risedronate is an orally administered pyridinyl bisphosphonate that is 36 times more potent than pamidronate and 72 times more potent than clodronate. Four randomized, double-blind trials have been carried out in patients with postmenopausal osteoporosis. In 2 of these studies, vertebral fracture incidence was reduced by a daily dose of 5 mg risedronate by up to 65% and 49% relative to placebo after 1 and 3 years, respectively. In these trials, risedronate improved lumbar spine, femoral neck, and femoral trochanter bone mineral density (BMD) at 6 months. In addition, preclinical studies have shown that risedronate is more potent than pamidronate and clodronate in inhibiting adhesion of prostate cancer cells to bone and preventing tumor cell invasion. The incidence of osteoporosis in prostate cancer patients has been well established; therefore, it is advantageous to assess the efficacy of oral bisphosphonate therapy.

DETAILED DESCRIPTION:
OUTLINE: This is a randomized, placebo-controlled, double-blind, multicenter, 2 arm study.

The study population will consist of prostate cancer patients with metastatic bone disease for whom androgen-deprivation therapy is planned. After stratification based on the patient's age, performance status, and severity of metastatic disease, the patients will be randomized at a 1:1 ratio to the following treatment arms:

* Daily oral risedronate combined with androgen deprivation
* Daily oral placebo combined with androgen deprivation

Initial clinical evaluation will be performed during the 2-week screening period. While patients receive per-protocol treatment, study assessments will be performed every 4 weeks during the first 3 months, and every 12 weeks thereafter.

Performance Status: Eastern Cooperative Oncology Group (ECOG) 0 to 2

Life Expectancy: At least 12 weeks

Hematopoietic:

* Absolute neutrophil count (ANC) > 1,000/mm3
* Platelet count > 100,000/mm3
* international normalized ratio (INR) < 1.5 x upper limit of normal unless on therapeutic anticoagulation
* Partial thromboplastin time (PTT) < 1.5 x upper limit of normal unless on therapeutic anticoagulation

Hepatic:

* Bilirubin < 1.5 mg/dL
* Alanine transaminase (ALT) < 2.5 x upper limit of normal

Renal:

* Creatinine clearance of > 30 mL/min (by Cockcroft-Gault)

Cardiovascular:

* No significant history of uncontrolled cardiac disease (i.e., uncontrolled hypertension, unstable angina, and congestive heart failure).

Pulmonary:

* Not specified

Calcium:

* Corrected serum calcium = (4.0 g/dL - actual albumin g/dL)x 0.8 + serum calcium

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the prostate with metastatic bone disease (by CT, MRI or bone scan) with plans to start or be < 30 days from beginning androgen deprivation therapy. Patients with lymph node or visceral metastases only are not eligible
* Patients may receive palliative radiation therapy at the investigators discretion during the first 4 weeks of beginning protocol therapy.

Exclusion Criteria:

* No neuroendocrine, small cell or transitional cell cancer of the prostate No abnormal bone metabolism (i.e., Paget's disease, untreated hyperthyroidism, untreated hyperprolactinemia, untreated Cushing's disease).
* No use of calcitonin within 14 days before being registered for protocol therapy or any previous use of bisphosphonates.
* No major surgery within 4 weeks of registration to protocol therapy.
* No adjuvant chemotherapy within 6 months of registration to protocol therapy.
* No previous chemotherapy for metastatic disease.
* No hormonal therapy in the adjuvant setting within 12 months of registration to protocol therapy; previous hormonal therapy must not have exceeded 6 months.
* No prior history of malignancy in the past 5 years with the exception of basal cell and squamous cell carcinoma of the skin.
* No history of allergy or drug reactions to bisphosphonates.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2003-10; Primary Completion 2008-02 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Sweeney, M.B.B.S., Study Chair — Hoosier Oncology Group, LLC
Locations (45):
- United States (31):
  - Center for Urological Research, La Mesa, California
  - San Bernadino Urological Associates, San Bernardino, California
  - Grove Hill Medical Center Urology, New Britain, Connecticut
  - Innovative Surgical Resources, Tampa, Florida
  - Medical & Surgical Specialists, LLC, Galesburg, Illinois
  - Peoria Urological Associates, Peoria, Illinois
  - Oncology Hematology Associates of SW Indiana, Evansville, Indiana
  - Center for Cancer Care at Goshen Health System, Goshen, Indiana
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Quality Cancer Center (MCGOP), Indianapolis, Indiana
  - Urology of Indiana, LLC, Indianapolis, Indiana
  - Urology Associates, Muncie, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Urologic Surgery Associates, Baltimore, Maryland
  - Drs. Werner, Murdock and Francis PA Urology Associates, Greenbelt, Maryland
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Kansas City Urology Care, Kansas City, Missouri
  - Siteman Cancer Center, St Louis, Missouri
  - Nevada Urology, Reno, Nevada
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Lawrenceville Urology, Trenton, New Jersey
  - Accumed Research Associates, Garden City, New York
  - Staten Island Urological Research, P.C., Staten Island, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Oregon Urology Specialists, Springfield, Oregon
  - Urological Associates of Lancaster, Lancaster, Pennsylvania
  - Triangle Urological Group, Pittsburgh, Pennsylvania
  - Salt Lake Research, Salt Lake City, Utah
  - David Reed, M.D., Seattle, Washington
  - Madigan Army Medical Center Urology Service, Tacoma, Washington
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
- Canada (14):
  - Southern Interior Medical Research, Inc., Kelowna, British Columbia
  - Andreou Research, Surrey, British Columbia
  - Dr. G. Steinhoff Clinical Research, Victoria, British Columbia
  - Dr. Allan Patrick Professional Corporation, Fredericton, New Brunswick
  - Male/Female Health and Research, Barrie, Ontario
  - Burlington Professional Centre, Burlington, Ontario
  - Urology Resource Centre, Burlington, Ontario
  - Hamilton District Urology Research Center, Hamilton, Ontario
  - Centre for Advanced Urological Research, Kingston, Ontario
  - London Region Cancer Program, London, Ontario
  - MOR Urology, Inc., Newmarket, Ontario
  - Male Health Centres, Oakville, Ontario
  - Scarborough General Hospital, Medical Mall, Scarborough Village, Ontario
  - University Health Network - Princess Margaret Division, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] C. Sweeney, W. M. Dugan II, R. Dreicer, F. Chu, G. Parks, K. Baker, D. Reed, K. Jansz, J. Zadra, C. T. Yiannoutsos. J Clin Oncol 28, 2010 (suppl; abstr e15000)
- [Derived] Jakob T, Tesfamariam YM, Macherey S, Kuhr K, Adams A, Monsef I, Heidenreich A, Skoetz N. Bisphosphonates or RANK-ligand-inhibitors for men with prostate cancer and bone metastases: a network meta-analysis. Cochrane Database Syst Rev. 2020 Dec 3;12(12):CD013020. doi: 10.1002/14651858.CD013020.pub2. PMID 33270906
- [Derived] Hahn NM, Yiannoutsos CT, Kirkpatrick K, Sharma J, Sweeney CJ. Failure to suppress markers of bone turnover on first-line hormone therapy for metastatic prostate cancer is associated with shorter time to skeletal-related event. Clin Genitourin Cancer. 2014 Feb;12(1):33-40.e4. doi: 10.1016/j.clgc.2013.07.002. Epub 2013 Oct 12. PMID 24126237

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Target patients were men with castrate resistant prostate cancer for whom androgen-deprivation therapy was planned. Patients were enrolled at multiple outpatient oncology clinics and urological practices in the United States and Canada. Recruitment period was December 2003 and August 2005.
Pre-assignment Details: 1:1 stratification was based on patient's age, performance status and severity of metastatic disease. Initial clinical evaluation was performed during the 2-week screening period. Both arms received at least 500 mg/day oral calcium carbonate and 400 IU of vitamin D.
Period: Overall Study
Arm/Group | Risedronate | Placebo
Started | 32 | 31
Completed | 32 | 31
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Risedronate | Placebo | Total
Number analyzed (Participants) | 32 | 31 | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 16
  >=65 years | 24 | 23 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.2 (9.5) | 70.2 (8.4) | 70.2 (8.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 32 | 31 | 63
Previous Adjuvant Hormone Therapy [Number; unit: participants]
  Yes | 2 | 5 | 7
  No | 30 | 26 | 56
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) from 0-5 that describes a patient's level of functioning where 0=Fully active, able to carry on all pre-disease performance without restriction and 5=Dead:
  participants
    ECOG 0 | 26 | 19 | 45
    ECOG 1 | 4 | 10 | 14
    ECOG 2 | 2 | 2 | 4
Disease Extent [Number; unit: participants] — Minimal disease was defined as metastases limited to the pelvic and axial skeleton.
  Extensive disease was defined as metastases involving the appendicular skeleton or visceral metastases
  participants
    Minimal Disease | 11 | 11 | 22
    Extensive Disease | 21 | 20 | 41
Comorbidity Score [Number; unit: participants] — Comorbidity Scores were determined using the Adult Comorbidity Evaluation-27 Index (ACE-27). The ACE-27 grades 27 cogent comorbid ailments on a scale from 0-3 where 0=None, 1=Mild, 2=Moderate, 3=Severe.
  The highest ranked comorbid ailment determines the overall comorbidity score.
  The data reported in this table represents the data that was collected before the termination of the study.
  participants
    None | 6 | 3 | 9
    Mild | 7 | 11 | 18
    Moderate | 12 | 11 | 23
    Severe | 3 | 5 | 8

OUTCOME MEASURES:

1. Primary Outcome: Numbers of SRE or Death Occurred Cumulatively
Description: Number of participants experiencing a SRE(skeletal-related event) or death occurred, cumulative from each arm ( a daily oral dose of 30 mg risedronate, or placebo)
Time Frame: 36 months
Measure: Number; unit: participants
Groups:
- Risedronate Arm: Daily oral risedronate combined with androgen deprivation
  Risedronate: Daily oral risedronate combined with androgen deprivation
Arm/Group | Risedronate Arm | Placebo Arm
Number analyzed (Participants) | 32 | 31
participants | 11 | 13
Statistical Analysis 1: Comparison: Risedronate Arm vs Placebo Arm; Test type: Superiority or Other; p = 0.3, Regression, Cox; Hazard Ratio (HR) = 2.08, 95% CI 2-sided [0.51 to 8.40]

2. Secondary Outcome: Rate of Patients Archiving a PSA (Prostate Specific Antigen) Nadir < 0.2 ng/mL
Time Frame: 36 months
Measure: Number; unit: percentage of participants
Arm/Group | Risedronate Arm | Placebo Arm
Number analyzed (Participants) | 32 | 31
percentage of participants | 50 | 29
Statistical Analysis 1: Comparison: Risedronate Arm vs Placebo Arm; Test type: Superiority or Other; p = 0.12, univariate analysis

3. Secondary Outcome: Time to Development of Hormone Refractory Disease
Time Frame: 36 months
Population: No data were collected for this Outcome Measure due to low accrual and subsequent study termination.
Arm/Group | Risedronate Arm | Placebo Arm
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Bone Turnover Marker Changes -- Urine Total Deoxypyridinoline (DPD)
Description: Urine total DPD median in response to treatment on both study arms at week 24. compare median from baseline and week 24.
  Deoxypyridinoline (DPD) is measured in hydrolyzed urine samples using high-performance liquid chromatography technique. After extraction of the cross-links and elimination of the urine impurities by a Bio-Rad SPE cartridge (Bio-Rad Laboratories, Hercules, CA), total DPD is eluted from reverse-phase high-performance liquid chromatography by ion pair chromatography with isocratic elution.
  The compounds are detected as a result of their natural fluorescence with a fluorescence detector
Time Frame: 24 weeks
Population: Number of Participants Analyzed reflects participants who had data available prior to study termination.
Measure: Median (Standard Deviation); unit: nmol/mmol creatinine
Arm/Group | Risedronate Arm | Placebo Arm
Number analyzed (Participants) | 22 | 22
nmol/mmol creatinine
  week 24 | 6.91 (4.17) | 12.62 (13.59)
  baseline | 8.83 (20.53) | 10.12 (31.83)
Statistical Analysis 1: Comparison: Risedronate Arm vs Placebo Arm; Test type: Superiority or Other; p < 0.001, Kruskal-Wallis

5. Secondary Outcome: Three- Year Survival Rate
Time Frame: 36 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Risedronate | Placebo
Number analyzed (Participants) | 32 | 31
percentage of participants | 72.5 [55.1 to 89.9] | 71.5 [51.5 to 91.5]

6. Secondary Outcome: Bone Turnover Marker Changes-- Urine N-telopeptide (NTX) Median
Description: Urine N-telopeptide (NTX) median changes between baseline and week 24. The assays are performed with the NTx Reagent Pack kit from Ortho-Clinical Diagnostics (Ortho-Clinical Diagnostics/Johnson & Johnson, Amersham, UK), which is a kit designed for the quantitative determination of N-terminal telopeptide (NTx) in human urine on the automated Vitros Immunodiagnostic System ECi (Ortho-Clinical Diagnostics/Johnson & Johnson, Amersham, UK). A competitive immunoassay technique is used. This depends on competition between NTx present in the sample and a synthetic NTx peptide coated on the wells for binding by a horseradish peroxidase (HRP)-labeled antibody conjugate (mouse monoclonal anti-NTx). The conjugate is captured by the peptide coated on the wells; unbound materials are removed by washing.
  The bound HRP conjugate is measured by a luminescent reaction.
Time Frame: 24 week
Population: Number of Participants Analyzed reflects participants who had data available prior to study termination.
Measure: Median (Standard Deviation); unit: nmol BCE/mmol creatinine
Arm/Group | Risedronate Arm | Placebo Arm
Number analyzed (Participants) | 20 | 19
nmol BCE/mmol creatinine
  at 24 week | 20.63 (9.15) | 62.95 (151.67)
  baseline | 41.33 (325.87) | 48.08 (691.70)
Statistical Analysis 1: Comparison: Risedronate Arm vs Placebo Arm; Test type: Superiority or Other; p < 0.001, Kruskal-Wallis

7. Secondary Outcome: Bone Turnover Marker Changes-- Serum BAP
Description: Serum BAP median changes between baseline and week 24. The Ostase assays are performed with an access immunoassay system, which is an assay of serum samples that provides a quantitative measurement of bone alkaline phosphatase (BAP). A mouse monoclonal antibody specific to BAP is added to a re-action vessel with paramagnetic particles coated with goat antimouse polyclonalantibody.Calibrators,controls,andsamplescontainingBAP are added to the coated particles and bind to the anti-BAP monoclonal antibody. After the formation of a solid phase/capture antibody/BAP complex, separation in a magnetic field and washing remove materials not bound to the solid phase. A chemiluminescent substrate, LumiPhos 530, is added to the reaction vessel, and light generated by the reaction is measured with a luminometer. The light production is directly proportional to the concentration of BAP in the sample. The amount of analyte in thesample is determined from a stored multipoint calibration curve
Time Frame: 24 week
Population: Number of Participants Analyzed reflects participants who had data available prior to study termination.
Measure: Median (Standard Deviation); unit: ng/mL
Arm/Group | Risedronate Arm | Placebo Arm
Number analyzed (Participants) | 19 | 17
ng/mL
  24 week | 9.5 (4.59) | 13.16 (54.62)
  baseline | 20.95 (229.68) | 19.50 (272.98)
Statistical Analysis 1: Comparison: Risedronate Arm vs Placebo Arm; Test type: Superiority or Other; p = 0.010, Kruskal-Wallis

8. Secondary Outcome: Bone Turnover Marker Changes-- Serum Osteocalcin (OC)
Description: Serum Osteocalcin (OC) medians between baseline and 24 weeks areperformed with the Elecsys 2010 automated analyzer, which uses an electrochemiluminescence immunoassay technique for the in vitro quantitative determination of serum total osteocalcin in humanserum. The assay uses a sandwich test principle in which afirst biotinylated monoclonal antibody recognizing N-MID osteocalcin and a second monoclonal antibody against N-MID osteocalcin labeled with ruthenium are incubated with 20mL of serum. After a first incubation, streptavidin-coated microparticles are added for a second incubation, and the complex becomes bound to the solid phase by interaction of biotin and streptavidin.These microparticles are then magnetically captured onto the surface of an electrode. Application of a voltage on this electrode induces chemiluminescent emission, which is measured by a photomultiplierand compared with a calibration curve that is generated in aninstrument-specific manner by 2-point calibration.
Time Frame: 24 week
Population: Number of Participants Analyzed reflects participants who had data available prior to study termination.
Measure: Median (Standard Deviation); unit: ug/L
Arm/Group | Risedronate Arm | Placebo Arm
Number analyzed (Participants) | 19 | 18
ug/L
  at 24 week | 11.88 (14.94) | 27.35 (57.43)
  baseline | 20.08 (38.36) | 18.24 (43.06)
Statistical Analysis 1: Comparison: Risedronate Arm vs Placebo Arm; Test type: Superiority or Other; p < 0.001, Kruskal-Wallis

ADVERSE EVENTS:
Time Frame: 36 Months
Arm/Group | Placebo | Risedronate
Serious Adverse Events (participants affected / at risk) | 5/31 | 8/32
Other Adverse Events (participants affected / at risk) | 26/31 | 29/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=31) | Risedronate (N=32)
CARDIAC GENERAL - OTHER (Cardiac disorders) | 0 (0) | 1 (1)
CARDIAC ISCHEMIA/INFARCTION (Cardiac disorders) | 2 (2) | 0 (0)
CONDUCTION ABNORMALITY/ATRIOVENTRICULAR HEART BLOCK / AV BLOCK-THIRD DEGREE (COMPLETE AV BLOCK) (Cardiac disorders) | 0 (0) | 1 (1)
CYSTITIS (Renal and urinary disorders) | 0 (0) | 1 (1)
DEHYDRATION (Gastrointestinal disorders) | 0 (0) | 2 (2)
HEMOLYSIS (E.G., IMMUNE HEMOLYTIC ANEMIA, DRUG-RELATED HEMOLYSIS) (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
INFECTION WITH UNKNOWN ANC / LUNG (PNEUMONIA) (Infections and infestations) | 1 (1) | 0 (0)
INFECTION WITH UNKNOWN ANC / URINARY TRACT NOS (Infections and infestations) | 1 (1) | 0 (0)
INR (INTERNATIONAL NORMALIZED RATIO OF PROTHROMBIN TIME) (Surgical and medical procedures) | 0 (0) | 1 (1)
LEFT VENTRICULAR SYSTOLIC DYSFUNCTION (Cardiac disorders) | 1 (1) | 0 (0)
MUSCLE WEAKNESS, GENERALIZED OR SPECIFIC AREA (NOT DUE TO NEUROPATHY) / WHOLE BODY/GENERALIZED (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PAIN / ABDOMEN NOS (Gastrointestinal disorders) | 1 (1) | 0 (0)
PAIN / PAIN NOS (General disorders) | 0 (0) | 1 (1)
PERFORATION, GU / KIDNEY (Renal and urinary disorders) | 1 (1) | 0 (0)
PLATELETS (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
PULMONARY FIBROSIS (RADIOGRAPHIC CHANGES) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
RENAL FAILURE (Renal and urinary disorders) | 1 (1) | 0 (0)
SODIUM, SERUM-LOW (HYPONATREMIA) (Investigations) | 0 (0) | 1 (1)
STRICTURE/STENOSIS (INCLUDING ANASTOMOTIC), GI / BILIARY TREE (Gastrointestinal disorders) | 1 (1) | 0 (0)
SUPRAVENTRICULAR AND NODAL ARRHYTHMIA / ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 1 (1)
THROMBOSIS/THROMBUS/EMBOLISM (Vascular disorders) | 2 (2) | 0 (0)
VESSEL INJURY-ARTERY / AORTA (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=31) | Risedronate (N=32)
ALT, SGPT (SERUM GLUTAMIC PYRUVIC TRANSAMINASE) (Investigations) | 2 (3) | 0 (0)
ANOREXIA (Gastrointestinal disorders) | 1 (1) | 3 (3)
ARTHRITIS (NON-SEPTIC) (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
AST, SGOT(SERUM GLUTAMIC OXALOACETIC TRANSAMINASE) (Investigations) | 1 (2) | 0 (0)
BILIRUBIN (HYPERBILIRUBINEMIA) (Investigations) | 1 (2) | 0 (0)
BRONCHOSPASM, WHEEZING (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
BRUISING (IN ABSENCE OF GRADE 3 OR 4 THROMBOCYTOPENIA) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
BURN (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
CARDIAC GENERAL - OTHER (Cardiac disorders) | 1 (1) | 0 (0)
CATARACT (Eye disorders) | 0 (0) | 1 (1)
CERVICAL SPINE-RANGE OF MOTION (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
CHOLESTEROL, SERUM-HIGH (HYPERCHOLESTREMIA) (Investigations) | 1 (1) | 1 (1)
CONFUSION (Nervous system disorders) | 1 (1) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 8 (8) | 8 (9)
CONSTITUTIONAL SYMPTOMS - OTHER (General disorders) | 6 (6) | 4 (9)
COUGH (Respiratory, thoracic and mediastinal disorders) | 5 (7) | 4 (5)
CREATININE (Investigations) | 1 (1) | 0 (0)
DERMATOLOGY/SKIN - OTHER (Skin and subcutaneous tissue disorders) | 5 (5) | 3 (5)
DIARRHEA (Gastrointestinal disorders) | 3 (3) | 5 (8)
DISTENSION/BLOATING, ABDOMINAL (Gastrointestinal disorders) | 1 (1) | 1 (1)
DIZZINESS (Nervous system disorders) | 2 (2) | 2 (2)
DRY MOUTH/SALIVARY GLAND (XEROSTOMIA) (Gastrointestinal disorders) | 3 (3) | 0 (0)
DRY SKIN (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
DYSPHAGIA (DIFFICULTY SWALLOWING) (Gastrointestinal disorders) | 0 (0) | 1 (1)
DYSPNEA (SHORTNESS OF BREATH) (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 4 (4)
EDEMA: LIMB (Blood and lymphatic system disorders) | 5 (6) | 5 (6)
ENDOCRINE - OTHER (Endocrine disorders) | 1 (1) | 0 (0)
ERECTILE DYSFUNCTION (Reproductive system and breast disorders) | 1 (1) | 0 (0)
EXTREMITY-LOWER (GAIT/WALKING) (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
EXTREMITY-UPPER (FUNCTION) (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
FATIGUE (ASTHENIA, LETHARGY, MALAISE) (General disorders) | 13 (19) | 12 (15)
FEVER (IN THE ABSENCE OF NEUTROPENIA, WHERE NEUTROPENIA IS DEFINED AS ANC <1.0 X 10E9/L) (General disorders) | 1 (1) | 0 (0)
FLUSHING (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
FRACTURE (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
GASTRITIS (INCLUDING BILE REFLUX GASTRITIS) (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTROINTESTINAL - OTHER (Gastrointestinal disorders) | 2 (2) | 4 (6)
GLUCOSE, SERUM-HIGH (HYPERGLYCEMIA) (Investigations) | 3 (6) | 0 (0)
GYNECOMASTIA (Reproductive system and breast disorders) | 1 (1) | 1 (1)
HAIR LOSS/ALOPECIA (SCALP OR BODY) (Skin and subcutaneous tissue disorders) | 1 (2) | 2 (2)
HEARTBURN/DYSPEPSIA (Gastrointestinal disorders) | 4 (4) | 6 (6)
HEMOGLOBIN (Blood and lymphatic system disorders) | 3 (3) | 2 (2)
HEMOLYSIS (E.G., IMMUNE HEMOLYTIC ANEMIA, DRUG-RELATED HEMOLYSIS) (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
HEMORRHAGE, GU / URINARY NOS (Renal and urinary disorders) | 1 (1) | 0 (0)
HEMORRHAGE, PULMONARY/UPPER RESPIRATORY / NOSE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
HOT FLASHES/FLUSHES (Endocrine disorders) | 16 (17) | 16 (20)
HYPERTENSION (Cardiac disorders) | 5 (6) | 1 (1)
HYPOTENSION (Cardiac disorders) | 0 (0) | 1 (1)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
INCONTINENCE, URINARY (Renal and urinary disorders) | 0 (0) | 1 (1)
INFECTION WITH GRADE 3 OR 4 NEUTROPHILS (ANC <1.0 X 10E9/L) / MIDDLE EAR (OTITIS MEDIA) (Infections and infestations) | 0 (0) | 1 (1)
INFECTION - OTHER (Infections and infestations) | 1 (1) | 2 (2)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / BLADDER (URINARY) (Infections and infestations) | 0 (0) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / JOINT (Infections and infestations) | 1 (1) | 0 (0)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / LUNG (PNEUMONIA) (Infections and infestations) | 1 (1) | 0 (0)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / NERVE-PERIPHERAL (Infections and infestations) | 1 (1) | 0 (0)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / PENIS (Infections and infestations) | 1 (1) | 0 (0)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / SKIN (CELLULITIS) (Infections and infestations) | 1 (1) | 0 (0)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / UPPER AIRWAY NOS (Infections and infestations) | 1 (1) | 0 (0)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / URINARY TRACT NOS (Infections and infestations) | 0 (0) | 1 (1)
INFECTION WITH UNKNOWN ANC / LUNG (PNEUMONIA) (Infections and infestations) | 1 (1) | 1 (1)
INFECTION WITH UNKNOWN ANC / UNGUAL (NAILS) (Infections and infestations) | 1 (1) | 0 (0)
INFECTION WITH UNKNOWN ANC / URINARY TRACT NOS (Infections and infestations) | 0 (0) | 1 (1)
INFECTION WITH UNKNOWN ANC / WOUND (Infections and infestations) | 1 (1) | 0 (0)
INJECTION SITE REACTION/EXTRAVASATION CHANGES (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
INSOMNIA (General disorders) | 6 (7) | 5 (5)
JOINT-EFFUSION (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
JOINT-FUNCTION (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (1)
LEAK (INCLUDING ANASTOMOTIC), GU / URETHRA (Renal and urinary disorders) | 0 (0) | 1 (1)
LUMBAR SPINE-RANGE OF MOTION (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
MOOD ALTERATION / AGITATION (Psychiatric disorders) | 1 (1) | 0 (0)
MOOD ALTERATION / ANXIETY (Psychiatric disorders) | 3 (3) | 0 (0)
MOOD ALTERATION / DEPRESSION (Psychiatric disorders) | 5 (5) | 3 (3)
MUSCLE WEAKNESS, GENERALIZED OR SPECIFIC AREA (NOT DUE TO NEUROPATHY) / EXTREMITY-LOWER (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
MUSCLE WEAKNESS, GENERALIZED OR SPECIFIC AREA (NOT DUE TO NEUROPATHY) / EXTREMITY-UPPER (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MUSCLE WEAKNESS, GENERALIZED OR SPECIFIC AREA (NOT DUE TO NEUROPATHY) / RIGHT-SIDED (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MUSCLE WEAKNESS, GENERALIZED OR SPECIFIC AREA (NOT DUE TO NEUROPATHY) / WHOLE BODY/GENERALIZED (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
MUSCULOSKELETAL/SOFT TISSUE - OTHER (Musculoskeletal and connective tissue disorders) | 3 (4) | 6 (11)
NAIL CHANGES (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
NASAL CAVITY/PARANASAL SINUS REACTIONS (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 4 (5) | 5 (6)
NEUROLOGY - OTHER (Nervous system disorders) | 2 (2) | 0 (0)
NEUROPATHY: CRANIAL / CN VII MOTOR-FACE; SENSORY-TASTE (Nervous system disorders) | 1 (1) | 0 (0)
NEUROPATHY: MOTOR (Nervous system disorders) | 0 (0) | 1 (1)
NEUROPATHY: SENSORY (Nervous system disorders) | 6 (9) | 6 (8)
OBESITY (General disorders) | 1 (1) | 0 (0)
OBSTRUCTION, GU / URETER (Renal and urinary disorders) | 1 (1) | 0 (0)
OCULAR/VISUAL - OTHER (Eye disorders) | 1 (1) | 1 (1)
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTITIS, MIDDLE EAR (NON-INFECTIOUS) (Ear and labyrinth disorders) | 0 (0) | 1 (1)
PAIN / ABDOMEN NOS (Gastrointestinal disorders) | 1 (1) | 0 (0)
PAIN / BACK (General disorders) | 6 (7) | 10 (12)
PAIN / BONE (Musculoskeletal and connective tissue disorders) | 4 (6) | 1 (1)
PAIN / BREAST (Reproductive system and breast disorders) | 0 (0) | 1 (1)
PAIN / EXTREMITY-LIMB (Musculoskeletal and connective tissue disorders) | 4 (5) | 5 (8)
PAIN / HEAD/HEADACHE (General disorders) | 1 (1) | 2 (2)
PAIN / JOINT (Musculoskeletal and connective tissue disorders) | 6 (9) | 5 (10)
PAIN / MUSCLE (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
PAIN / NECK (General disorders) | 2 (2) | 3 (3)
PAIN / PAIN NOS (General disorders) | 0 (0) | 2 (3)
PAIN / PENIS (Reproductive system and breast disorders) | 0 (0) | 1 (1)
PAIN / SCROTUM (Reproductive system and breast disorders) | 1 (1) | 0 (0)
PAIN / TESTICLE (Reproductive system and breast disorders) | 2 (2) | 0 (0)
PAIN - OTHER (General disorders) | 1 (1) | 3 (6)
PLATELETS (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
PRURITUS/ITCHING (Skin and subcutaneous tissue disorders) | 5 (5) | 2 (3)
PULMONARY/UPPER RESPIRATORY - OTHER (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
RASH/DESQUAMATION (Skin and subcutaneous tissue disorders) | 3 (4) | 2 (2)
RASH: ACNE/ACNEIFORM (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
RENAL/GENITOURINARY - OTHER (Renal and urinary disorders) | 3 (6) | 3 (3)
RESTRICTIVE CARDIOMYOPATHY (Cardiac disorders) | 0 (0) | 1 (2)
RIGHT FOREARM LESION (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
SECONDARY MALIGNANCY - POSSIBLY RELATED TO CANCER TREATMENT (SPECIFY, __) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
SEIZURE (Nervous system disorders) | 1 (1) | 0 (0)
SODIUM, SERUM-LOW (HYPONATREMIA) (Investigations) | 1 (1) | 0 (0)
SUPRAVENTRICULAR AND NODAL ARRHYTHMIA / SINUS BRADYCARDIA (Cardiac disorders) | 1 (1) | 0 (0)
SWEATING (DIAPHORESIS) (General disorders) | 3 (4) | 1 (1)
SYNCOPE (FAINTING) (Nervous system disorders) | 1 (1) | 0 (0)
THROMBOSIS/EMBOLISM (VASCULAR ACCESS-RELATED) (Vascular disorders) | 1 (1) | 0 (0)
THROMBOSIS/THROMBUS/EMBOLISM (Vascular disorders) | 0 (0) | 2 (2)
UPPER RESPIRATORY INFECTION (Infections and infestations) | 1 (1) | 1 (1)
URINARY FREQUENCY/URGENCY (Renal and urinary disorders) | 7 (8) | 7 (8)
URINARY RETENTION (INCLUDING NEUROGENIC BLADDER) (Renal and urinary disorders) | 1 (1) | 1 (1)
VOICE CHANGES/DYSARTHRIA (E.G., HOARSENESS, LOSS OR ALTERATION IN VOICE, LARYNGITIS) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
VOMITING (Gastrointestinal disorders) | 2 (3) | 2 (2)
WATERY EYE (EPIPHORA, TEARING) (Eye disorders) | 0 (0) | 1 (1)
WEIGHT GAIN (General disorders) | 1 (3) | 0 (0)
WEIGHT LOSS (General disorders) | 1 (1) | 2 (2)
WOUND COMPLICATION, NON-INFECTIOUS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No